CLINICAL TRIAL: NCT00721669
Title: A Phase I Dose-Escalation Study of IMGN388 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN388
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Solid Tumor
Keywords: solid tumor

INTERVENTIONS:
Drug: IMGN388 — IMGN388 is a human IgG1 anti-integrin antibody conjugated to the maytansinoid, DM4.

SUMMARY:
Primary objective is to evaluate the safety and PK of IMGN388

DETAILED DESCRIPTION:
The secondary objectives are to assess the pharmacodynamics, immunogenicity, and tumor response of IMGN388 administered as an IV infusion once every three weeks in patients with solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Male or female age greater than 18 years
* Signed informed consent(s): Patients must provide informed consent for study participation prior to performing any study-specific procedures
* Histologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Specifically for the dose expansion phase, enrollment will be limited to patients with αv integrin positive melanomas or carcinomas of breast, lung, or ovary. Patients must also have confirmation of αv integrin expression performed prior to enrollment by immunohistochemical assessment for αv integrin on archived or if not available, freshly collected tumor biopsy samples. αv integrin positive tumors are defined as having a staining intensity of at least 2+ and a staining uniformity of heterogeneous (25 - 75% of tumor cells stain positively for αv integrin) or homogeneous staining (>75% of tumor cells are positive for αv integrin) of tumor cells when evaluated by immunohistochemistry .
* Evidence of measurable or evaluable metastatic disease at baseline
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of less than or equal to 2
* Adequate bone marrow, liver, and renal function at the time of first dose of study agent, as described below:
* Hemoglobin greater than or equal to 9.0 g/dL (5.6 mmol/L; 90 g/L) without transfusion dependency
* Absolute neutrophil count (ANC)greater than or equal to 1.5 x 109/L (1500/mm3) without hematopoietic cytokine support
* Platelets greater than or equal to 100,000 x 109/L (100,000/mm3) without transfusion dependency
* Coagulation [prothrombin time (PT) or international normalized ratio (INR) and activated partial prothrombin time (aPTT)] ≤ 1.25 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN if no liver metastasis; ≤ 5 x ULN if liver metastasis
* Total Bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN
* Female patients must be postmenopausal (at least 12 months since last menses), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before study entry, for the duration of study participation, and for three months after the last infusion of study agent and must have a negative urine or serum pregnancy test within 1 week before beginning treatment on this study and at all specified timepoints throughout the study. Men must be sterilized or agree to use a double-barrier method of birth control and must agree to not donate sperm during the study and for three months after the last infusion of study agent.
* Able to adhere to study visit schedule and all protocol requirements
* The anticipated life expectancy is such that the patient is expected to be able to participate for the duration of the study

Exclusion Criteria:

Patients meeting any of the following criteria may not be enrolled in the study:

* Residual toxicities resulting from previous therapy that are ≥ Grade 1
* Neuropathy of > Grade 1
* History of uveitis within 6 months of first dose of study agent or presenting with uveitis at baseline
* Concomitant or prior malignancy (other than the one under study) except adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Patients with solid tumors with history of active bleeding
* Treatment with systemic cancer therapy, radiotherapy or any investigational agent within 4 weeks or five half-lives (whichever is longer) of first dose of study agent
* Known allergies or clinically important reactions to human proteins or to therapeutic antibodies
* Major surgery within 4 weeks of first dose of study agent, or planning to have surgery (except for minor surgical procedures) during the study, or planned major surgery within 8 weeks after the last dose of study agent
* Serious concurrent illness (medical or psychiatric), altered mental status (e.g., dementia) or any uncontrolled medical condition (eg, uncontrolled diabetes), including the presence of laboratory abnormalities, that would place the patient at unacceptable risk by participating in the study or would confound the ability to interpret data from the study
* Uncontrolled infection, clinically important active infection within 4 weeks before the first dose of study agent, or currently receiving treatment for an infection
* Active angina pectoris or New York Heart Association (NYHA) Class III or IV heart disease. Cardiac disease characterized by significant ischemic coronary disease, significant arrhythmias, or congestive heart failure (greater than NYHA Class II) or myocardial infraction within the past 6 months
* Known or symptomatic central nervous system (CNS) metastases
* Known to be seropositive for human immunodeficiency virus (HIV), or active Hepatitis A, B, or C infection
* Any other concomitant anti-cancer treatment such as immunotherapy, biotherapy, radiotherapy, chemotherapy, investigative therapy, or high-dose steroids; however, low-dose steroids and Luteinizing Hormone Releasing Hormone (LHRH) at doses that have been stable for ≥ 14 days are permitted for patients with prostate cancer
* Any medical condition that, in the opinion of the investigator, may compromise the safety of the patient or their ability to receive study treatment
* Pregnant or lactating women

Patients will continue to be followed for short term follow-up and long term survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
evaluate the safety | during study
evaluate pharmacokinetics | during study

SECONDARY OUTCOMES:
assess the pharmacodynamics | during study
assess immunogenicity | during study
assess tumor response | during study

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee